CLINICAL TRIAL: NCT04135105
Title: Lexical Tone Perception in Tone Language speakers--a fMRI Study
Brief Title: Lexical Tone Perception in Tone language--a fMRI Study
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Kathy Y.S. LEE, Chief of Division of Speech Therapy, Chinese University of Hong Kong
Other Study IDs: Lexical tone perception(fMRI)
Record Dates: First submitted 2019-10-19; First posted 2019-10-22 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Lexical Tone; Neuroimaging; Chinese; Speech Perception
Keywords: Speech Perception; Neuroimaging; Lexical Tone; Chinese

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal hearing group: Right-handed, normal hearing, no reported neurological disorders
  Interventions: Other: Normal hearing group

INTERVENTIONS:
Other: Normal hearing group — Observational

SUMMARY:
Tone language refers to a language that uses fixed pitch pattern to distinguish words (Yip, 2002). Understanding the functional anatomy of the brain during lexical tone processing will provide useful hints for an effective intervention strategy such as brain stimulation. The present study investigate the cortical organisation of the brain in lexical tone perception of Cantonese speakers by the use of functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Tone language refers to a language that uses fixed pitch pattern to distinguish words (Yip, 2002). Cantonese is one of the main tone languages spoken by over 70 million around the world (Li et al.,1995; Adolfsson, 2010). Individuals with significant hearing impairment often present great difficulty in tone perception, affecting their understanding of words and hence, hamper their overall communication. The poor tone perception persists even with intensive auditory training coupled with advanced hearing technology such as cochlear implants.

Understanding the functional anatomy of the brain during lexical tone processing will provide useful hints for an effective intervention strategy such as brain stimulation. Researchers have been investigating the neural basis for tone perception in the past decades but failing to come to a consensus on the location of the brain that is responsible for lexical tone processing. The discrepant results may be due to the fact of the differences in subject selection (animals, healthy adults, brain-injured patients, tonal-language and non-tonal language speakers), testing materials and tasks employed (linguistic versus non-linguistic stimuli; dichotic listening versus discrimination and identification tasks) and outcome measurements (performance score, reaction time, accuracy rate, PET scan and fMRI).

Cortical organization, or brain mapping, refers to functional anatomy of the brain. The present study is the first study to systematically investigate the cortical organization of the brain in lexical tone perception of Cantonese speakers by the use of functional magnetic resonance imaging (fMRI). A comprehensive set of auditory stimuli specifically for investigating the different levels of lexical tone processing will be constructed. Native Cantonese speakers with normal hearing were recruited. They underwent fMRI while listening to the carefully designed auditory stimuli.

Once the cortical organization of lexical tone processing in Cantonese is identified, the valuable findings could be applied in further brain intervention procedures to tackle the long lasting, unresolved tone perception difficulty encountered by people with hearing impairment or other related disorders.

ELIGIBILITY:
Inclusion Criteria:

* native Cantonese speaker
* right-handed
* normal hearing
* no reported of neurological disorder

Exclusion Criteria:

* neurological disorder
* left-handed
* hearing impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruitment via University mass mail They were paid for their participations.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Activation areas in the brain that are responsible for lexical tone perception | 2015-2019
  To identify the activation area(s) in the brain that are responsible for lexical tone perception in normal hearing participants

SECONDARY OUTCOMES:
Accuracy rate | 2015-2019
  Accuracy rate of passive listening task
Reaction Time | 2015-2019
  reaction time of passive listening task

CONTACTS AND LOCATIONS:
Overall Officials: Yuet Sheung Lee, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided